CLINICAL TRIAL: NCT03198988
Title: Functionality and Accuracy of the smART System in Real-Life ICU Settings
Status: Terminated | Type: Interventional
Why Stopped: Due to the company's intent to conduct a new study under a different protocol with the smART+ System which is a more advanced version of the smART System.
Sponsor: ART Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CLT3_SY_P001
Record Dates: First submitted 2017-06-12; First posted 2017-06-26 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2021-07

CONDITIONS: Aspiration Pneumonia
MeSH Terms: conditions — Pneumonia, Aspiration

STUDY DESIGN:
Oversight: Unapproved Device: Yes

ARMS (1):
- General (Experimental): One arm study: smART Feeding Tube System.
  Interventions: Device: smART Feeding Tube System

INTERVENTIONS:
Device: smART Feeding Tube System — Replacing generic feeding tube with smART Feeding Tube System.

SUMMARY:
Total participants in the "Functionality and Accuracy of the smART System in Real-Life ICU Settings" are 10 participants - in the current Jefferson study site there were 8 participants and in the Sheba study site (identifier NCT03689985) there were 2 participants.

This study is conducted in order to validate the functionality and accuracy of the smART™ System in a real-life ICU setting. The smART™ Feeding Tube System is a novel system with nasogastric tube developed by ART Medical (Healthcare) Ltd, based on sensor-lined tubes that transmit real-time information to an external console. The smART™ feeding tube is equipped with reflux sensors which alert when gastric contents regurgitating into the esophagus. In addition, the smART™ feeding tube is equipped with sensors designed to provide information about the location of the tube thus assisting in reducing the incident of misplacement during first positioning. The smART™ feeding tube is also automatically and in real-time stops feeding if the feeding tube moves out of position during ongoing use or detect gastric content in esophagus. Furthermore, smART™ Feeding Tube System can guide operator to correctly re-position the tube. Lastly the smART™ Feeding Tube System is equipped with an anti-reflux mechanism and automatic Gastric Residual Volume (GRV).

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years or older
* Patient has already been admitted to ICU
* Patient requires enteral feeding
* Patients receiving Proton Pump Inhibitors (PPI) therapy
* Informed consent by independent physician and next of kin
* ICU ventilated patients

Exclusion Criteria:

* Patients with anomalies or diseases of the esophagus and or stomach.
* Patients with known sensitivities or allergies to any of the feeding tube materials
* Inability to place patient in semi-Fowler's position.
* Any clinically significant abnormality upon physical examination which may, in the opinion of the investigator, pose difficulty in inserting the feeding tube (e.g. cervical spine disorder)
* Pregnancy
* Recent abdominal surgery (less than 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- smART Feeding Tube System: The smART™ Feeding Tube System is a novel feeding tube developed by ART Healthcare Ltd. to overcome feeding tube displacement and reflux prevention and the complications associated with them. The smART Feeding Tube is equipped with sensors designed to provide information about the location of the tube tip relative to the lower esophageal sphincter as well as a balloon intended to aid in the prevention of aspiration due to reflux episodes.
Period: Overall Study
Arm/Group | smART Feeding Tube System
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | General
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 53.62 [18 to 120]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
  Israel | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants for Whom the System is Able to Accurately Guide and Ensure Correct Initial Feeding Tube Placement , Verified by X-ray
Time Frame: Enrollment visit
Measure: Count of Participants; unit: Participants
Arm/Group | General
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: Number of Tube "Out of Position" Alerts During Ongoing Use
Description: Any patient , in which the system alerted of tube out of position , the staff verified this according to the tube markings and if mispositioning occurred, this was documented the event in the CRF "out of position"
Time Frame: Enrollment day up to 7 days
Population: Number of events that system is able to detect tube movement during the study period .
Measure: Number; unit: Out of position alerts
Arm/Group | General
Number analyzed (Participants) | 9
Out of position alerts | 16

3. Primary Outcome: Number of Automatic System Generated Feeding Stops in Response to Tube Displacement.
Description: In order to prevent aspiration, the system software automatically pinches the feeding tube. Verification of the functionality of automatic feeding cessation when tube displacement is detected was done as part of the formal verification of the system
Time Frame: From insertion of feeding tube up to its removal , an average of 7 days.
Measure: Number; unit: Number of stops of feeding
Arm/Group | smART Feeding Tube System
Number analyzed (Participants) | 9
Number of stops of feeding | 16

4. Primary Outcome: Number of Major Reflux Event That Lead to Automatically Stops Feeding
Description: Overfeeding is the intolerance of the stomach to feeding material that causes reflux. There are two types of reflux events as defined by the system; minor-reflux and massive-reflux. Both types of reflux events are detected by the level of fluids interacting with the sensors, the severity is defined by gastric content reaching above the lower esophageal sphincter (LES):
  1. Minor reflux is defined as gastric content that did not pass the balloon located in the center of the esophagus.
  2. Massive reflux is defined as gastric content that reaches immediately above the balloon.
Time Frame: From insertion of feeding tube up to its removal , an average of 7 days.
Population: Each time the system detected massive reflux the system stop the feeding
Measure: Number; unit: Massive reflux episodes
Arm/Group | General
Number analyzed (Participants) | 9
Massive reflux episodes | 709

5. Primary Outcome: Average Duration of Balloon Inflation in Response to a Reflux Episode.
Description: Massive reflux of gastric content can aspirate into the lungs and cause pneumonia. The system detects the reflux event and will (according to an algorithm) stop the feeding and or inflate a balloon and evacuate gastric residuals from the stomach to lower the risk of aspiration.
Time Frame: From insertion of feeding tube up to its removal , an average of 7 days.
Measure: Mean (Full Range); unit: Minutes
Arm/Group | General
Number analyzed (Participants) | 9
Minutes | 6.25 [0 to 87.81]

6. Secondary Outcome: Recording of Impedance Detected by the System and Correlation to Patient Positioning.
Description: Positions changes were correlated to reflux events captured by the system console. Any position change of the patient was captured by the video camera located above the patient's bed.
Time Frame: From insertion of feeding tube up to its removal , an average of 7 days.
Measure: Mean (Full Range); unit: position changes
Arm/Group | General
Number analyzed (Participants) | 9
position changes | 46.19 [38.46 to 77.27]

7. Secondary Outcome: Number of Participant With Change in Ventilator Associated Pneumonia (VAP) and/or Acute Respiratory Distress Syndrome (ARDS) as a Measure of Effectiveness in Reducing Aspiration of Gastric Contents
Description: The first and the last X-ray images obtained for patients during the study were used to evaluate Ventilator Associated Pneumonia (VAP) and/or Acute respiratory distress syndrome (ARDS)
Time Frame: 56 - 168 hours per patient
Measure: Count of Participants; unit: Participants
Arm/Group | smART Feeding Tube System
Number analyzed (Participants) | 9
Participants
  Improvement in VAP/ARDS according to X-ray | 4
  No VAP/ cannot be estimated | 3
  No chance from first and last Xray images is seen | 2

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | General
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | General (N=10)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Hypothermia (General disorders) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
ARDS (Vascular disorders) | 1 (1)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ventricular bigeminy (Cardiac disorders) | 1 (1)
CHF (Cardiac disorders) | 1 (1)
Left femoral deep vein thrombosis (Vascular disorders) | 1 (1)
Febrile (General disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Colonic ileus (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT03198988/Prot_SAP_000.pdf